CLINICAL TRIAL: NCT04924491
Title: Randomized, Exploratory and Prospective Phase I/II Clinical Trial to Evaluate the Safety and Efficacy of the Transfusion of Autologous Treg Cells Obtained From Thymic Tissue in the Prevention of Rejection in Heart Transplant Children
Brief Title: Cell Therapy With Treg Cells Obtained From Thymic Tissue (thyTreg) to Prevent Rejection in Heart Transplant Children
Acronym: THYTECH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rafael Correa-Rocha (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Rafael Correa-Rocha, Group Leader, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THYTECH1-2018-005; 2024-519845-30 (EudraCT Number); 2018-003574-28 (Other: AEMPS)
Record Dates: First submitted 2021-04-30; First posted 2021-06-14 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-10

CONDITIONS: Heart Transplantation
Keywords: Cardiac Disease; Regulatory T cell; Immunomodulation; Tolerogenic protocol; Immunosuppressive Agents; Immunologic Factors
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10.000.000 thyTreg /kg (Experimental): Autologous thyTreg 10.000.000
  Interventions: Biological: Autologous thyTreg
- 20.000.000 thyTreg /kg (Experimental): Autologous thyTreg 20.000.000
  Interventions: Biological: Autologous thyTreg

INTERVENTIONS:
Biological: Autologous thyTreg — Treg lymphocytic cells, differentiated, autologous, of thymic tissue, expanded and stimulated with Interleukin (IL-) 2 (thyTreg)
  Other Names: thyTreg cells

SUMMARY:
The investigators developed a protocol to isolate Treg cells from thymic tissue (thyTreg) discarded in pediatric cardiac surgeries. After completing the pre-clinical studies, the investigators have initiated a phase I/II clinical trial to test the safety and efficacy of the adoptive transfer of autologous thyTreg to prevent rejection in heart transplant children.

Condition or disease: Heart Transplantation Intervention/treatment: Regulatory T Cell (Treg) Infusion

DETAILED DESCRIPTION:
Current transplant practice is far from guaranteeing the life expectancy of patients, particularly if the patients are children. THYTECH aims to revolutionize the field of clinical immunology developing a new approach to govern the regulatory skills of immune system, preventing graft rejection and opening a new frontier in the treatment of immune diseases.

Transfer of regulatory T cells (Treg) has acquired growing interest in the race to achieve indefinite transplant survival. Up to now, the use of Treg therapy to prevent solid graft rejection in humans has demonstrated that this therapy is safe, but the clinical efficacy is limited. The small Treg numbers that can be purified from peripheral blood along with the low survival and limited suppressive capacity of differentiated Tregs obtained from adults have probably compromised the efficacy of this therapy.

The investigators have developed an innovative approach to overcome current barriers and make Treg transfer a reality equipped to achieve indefinite graft survival. The major innovation of THYTECH is the employment of thymic tissue, the site of Treg generation, as a new source of Tregs to obtain massive amounts of thymus-derived Tregs (thyTreg) with very high purity (>95% of CD 25+ Foxp3+ cells) and improved survival and suppressive capacities. The investigators are recruiting patients in a clinical trial transferring autologous Tregs in heart-transplanted children to prevent graft rejection.

ELIGIBILITY:
Inclusion Criteria:

1. Patient under two years of age, who meets all the necessary requirements to undergo a heart transplant.
2. Patients without contraindication to immunosuppressive drugs.
3. Parents and/or guardians must be willing and able to understand the purpose and risks of the study and must sign the informed consent document

Exclusion Criteria:

1. Patients with DiGeorge Syndrome, since their thymic function is affected.
2. Human immunodeficiency virus positive serology
3. Epstein-Barr virus active infection
4. Patients hyperimmunized with cytotoxic anti-human leukocyte antigen antibodies
5. Patients with a history of previous malignancy
6. Patients who have participated in other intervention studies in the last month.
7. Patients who have received induction therapy with Basiliximab or Thymoglobulin.
8. Patients who have previously been thymectomized or transplanted.
9. Patients who have been diagnosed with severe autoimmune disease (celiac disease, autoimmune hypothyroidism, autoimmune diabetes)
10. Patients who will receive an asystole heart

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Repopulation of Treg cells in the patient, determined as the increase of Treg values in peripheral blood with respect to pre-transplant values or in comparison with a control cohort of non-treated patients. | 24 months

SECONDARY OUTCOMES:
Incidence of episodes of acute myocardial rejection (diagnosed by echocardiography) that require treatment in the 2 years post-transplant | 24 months
Number of Treg cells in peripheral blood | 24 months
Change in the number of naive and memory Treg cells, and the production/levels of interferon gamma and interleukins (IL-4, IL-17A and IL-10). | 24 months
Decrease of cell subsets related with rejection (CD8 T cells subsets, activated T cells, antibody-secreting B cells) during the post-transplant follow-up period. | 24 months
Overall patient survival rate at 24 months. | 24 months
Change on parameters of electrocardiogram (PR, QRS and corrected QT interval) of transplanted heart. | 24 months
Change on parameters of echocardiogram (mitral and tricuspid regurgitation; mitral and tissue mitral Doppler; and tricuspid and tissue tricuspid Doppler ) of transplanted heart. | 24 months
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE V4.03 criteria. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Correa-Rocha, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernaldo-de-Quiros E, Cozar B, Lopez-Esteban R, Clemente M, Gil-Jaurena JM, Pardo C, Pita A, Perez-Caballero R, Camino M, Gil N, Fernandez-Santos ME, Suarez S, Pion M, Martinez-Bonet M, Correa-Rocha R. A Novel GMP Protocol to Produce High-Quality Treg Cells From the Pediatric Thymic Tissue to Be Employed as Cellular Therapy. Front Immunol. 2022 May 16;13:893576. doi: 10.3389/fimmu.2022.893576. eCollection 2022. PMID 35651624